CLINICAL TRIAL: NCT07255599
Title: Tetrahydrobiopterin Responsiveness in Phenylketonuria Prediction With the 48-hour Loading Test and Genotype
Brief Title: Evaluation of BH4 Responsiveness in Our PKU Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Gadelkarim Mohamed, principal investigator, Sohag University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med--25-9-6MS
Record Dates: First submitted 2025-09-25; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GROUP 1 (Active Comparator): Sapropterin Dihydrochloride
  Interventions: Drug: Sapropterin Dihydrochloride (BH4, tetrahydrobiopterin)

INTERVENTIONS:
Drug: Sapropterin Dihydrochloride (BH4, tetrahydrobiopterin) — Patients were supplemented with phenylalanine a protein rich supplement based on milk protein, or an increase in natural protein intake) if phenylalanine was < 400 μmol/l. BH4 20 mg/kg was administered at T = 0 and T = 24. Blood samples were taken at T = 0, 8, 16, 24 and 48 h. Responsiveness was defined as ≥ 30% reduction in phenylalanine concentration at ≥ 1 time point.

SUMMARY:
This study aims to evaluate BH4 responsiveness in our PKU patients and to correlate BH4 responsiveness with their genotype

ELIGIBILITY:
Inclusion Criteria:

* Patients were supplemented with phenylalanine a protein rich supplement based on milk protein, or an increase in natural protein intake) if phenylalanine was < 400 μmol/l

Exclusion Criteria:

* if phenylalanine was less than 400 μmol/l

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
• Serum phenylealanine level in patients after given tetrahydrobiopterin | Blood samples were taken at Hour = 0, 8, 16, 24 and 48
  Patients were supplemented with phenylalanine a protein rich supplement based on milk protein, or an increase in natural protein intake) if phenylalanine was < 400 μmol/l. BH4 20 mg/kg was administered for 48 hours . Blood samples were taken at Hour = 0, 8, 16, 24 and 48 . Responsiveness was defined as ≥ 30% reduction in phenylalanine concentration at ≥ 1 time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided